CLINICAL TRIAL: NCT03369652
Title: Can Telephone Contact After Discharge Between Geriatrician, Clinical Pharmacist and General Practitioner About Medication Review in Hospital Improve the Medication in Older Patients? A Feasibility Study.
Brief Title: Telephone Contact Between Hospital and General Practitioner About Medication Review for Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lene V. Ravn-Nielsen, Pharmacist, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OP_468; 1704197 (Other Grant/Funding Number: Sundheds- og Ældreministeriet)
Record Dates: First submitted 2017-11-21; First posted 2017-12-12 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Older Patients; Medication Review; Cross-sectional Communication
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Medication history by pharmaconomist. Medication review by pharmacist, patient interview, and conference with physician in hospital, telephone contact to general practitioner after discharge, medication report sent to primary care.
  Interventions: Behavioral: Medication review
- Control (No Intervention): Medication history by pharmaconomist. Usual care by physicians.

INTERVENTIONS:
Behavioral: Medication review — Conducted by the pharmacist and discussed with hospital physician
  Arms: Intervention

SUMMARY:
In this trial, the feasibility of cooperation between clinical pharmacists and physicians by conducting a telephone follow-up conversation between the hospital geriatrician, the general practitioner and the clinical pharmacist is evaluated. During hospital stay the clinical pharmacist and the geriatrician will review older patients' medication and discuss the future treatment with the general practitioner after discharge by telephone or medico-technology.

The first part of the feasibility study will be a qualitative baseline measure of characteristics of the participants and work flow. The second part will be a pilot randomized controlled study where participants will be allocated to either usual care or medication review and follow up contact

ELIGIBILITY:
Inclusion Criteria:

* 5 drugs or more

Exclusion Criteria:

* Terminal illness
* Not able to speak and understand Danish

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in number of medications | At admission and at discharge
  Increase or decrease in number of medications from admission to discharge
Parts of the intervention completed | Day 1 after discharge
  In the intervention Group only, it is measured, how many of the elements of the intervention the patient actually have received
Changes in the Electronic Medication Profile (FMK) | 14 days after discharge
  How many changes have been Applied to the Electronic Medication Profile

SECONDARY OUTCOMES:
Number of readmissions | within 30 days after discharge
  Data from registers
Number of emergency visits | within 30 days after discharge
  Data from registers
Number of visits at general practitioner | within 30 days after discharge
  Data from registers
Patient satisfaction with the discharge | 14 days after discharge
  Measured by telephone interview
Changes in patient-experienced quality of life | At admission and 14 days after discharge
  Measured by telephone interview using the 5-item questionnaire EQ-5D, where each question can be answered on a 5-point Likert Scale ranging from "very high degree of problems" to "very low degree of problems"
Health care professionals satisfaction | 3 months after implementation
  Measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anton Pottegård, phd, Study Chair — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - Svendborg Sygehus, Svendborg

IPD SHARING:
Plan to Share IPD: No
No IPD are planned sharing